CLINICAL TRIAL: NCT05611112
Title: Problem-Solving Therapy for Patients With Chronic Disease and Poor Mental Well-being in General Practice
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Research Unit for General Practice, Aarhus University (Other); Danish Heart Foundation (Other); TrygFonden, Denmark (Industry); Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PST
Record Dates: First submitted 2022-10-28; First posted 2022-11-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Mental Health Impairment; Diabetes Type 2; Ischemic Heart Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster-randomised controlled trial with a one-year follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control group will have unrestricted access to care as usually provided. No restrictions are imposed on the general practitioners (GPs) regarding treatment of patients with mental health problems, as we are interested in assessing the added value of PST in routine clinical practice. In both groups, GPs are recommended to follow the current guidelines.
- Intervention (Experimental): Patients with type 2 diabetes and/or chronic ischemic heart disease are offered up to seven problem solving therapy sessions within a three-month period from inclusion. In both groups, GPs are recommended to follow the current guidelines.
  Interventions: Behavioral: Problem Solving Therapy

INTERVENTIONS:
Behavioral: Problem Solving Therapy — Problem Solving Therapy is a well-established evidence-based therapy form that is highly effective in patients with mental health issues. Initially, the patient makes a problem list and for each problem, possible solutions will be outlined. Considering pros and cons for each solution, the patient is asked to choose the one considered most appropriate. The patient is encouraged to put this solution into action and a follow-up consultation is planned.
  Arms: Intervention

SUMMARY:
In Denmark the vast majority of patients with chronic ischemic heart disease and/or type 2 diabetes are managed in general practice. 20% of the patients suffer from poor mental health.

Problem-solving therapy (PST) is a psychotherapeutic method that is proven effective in adults with poor mental health. PST can be provided in general practice.

The main objective of this study is to test effectiveness of providing PST to this group patients.

DETAILED DESCRIPTION:
20% of patients with type 2 diabetes and/or chronic ischemic heart disease have poor mental health. Since these patients are managed in general practice interventions targeting poor mental health in these patients should be delivered in here.

Problem-solving therapy (PST) is a well-established psychotherapeutic method that can be delivered by health care providers in general practice.

The main objective of this study is to test the effectiveness of delivering PST for patients with T2D and/or IHS who suffer from poor mental health. We hypothesize that the patients' mental health will be improved after treatment with PST.

Health care providers from 12 general practices are trained in PST and subsequently provide PST for patients with T2D and/or IHS and poor mental health.

Patients are recruited at the annual control visit for the chronic disease. All patients are screened for impaired mental health with the WHO-5 questionnaire. Patients with a score below 50 are offered PST.

The study is conducted as a stepped wedge cluster-randomised controlled trial with a one-year follow-up. In this design clusters are stepped wise exposed to the intervention. Initially all general practices are in the control group. After four months half of the recruited GPs attend the PST training programme and switch to performing the intervention. After an additional four months the remaining GPs are educated in PST and all GPs now perform the intervention. Both general practitioners and practise nurses will perform PST consultations.

The power calculation is based on:

* The primary outcome (PHQ-9 score at 6 and 12 months. The minimal clinical effect is 5 points)
* ICC is estimated to 0,05.

Based on these assumptions we will include 188 patients with IHS or/and T2D (we expect 25% overlap) to obtain a power of 90%.

ELIGIBILITY:
Inclusion Criteria:

* +18 years
* Diagnosed with ischemic heart disease and/or type 2 diabetes
* Poor mental health defined as WHO-5 well-being index <50 points

Exclusion Criteria:

* severe mental illness including psychotic disease and suicidal behaviour
* unable to read and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Mental health - Depression | 12 months
  Patient Health Questionnaire-9 (PHQ-9) at 12 months of follow-up

SECONDARY OUTCOMES:
Mental health - Anxiety | 12 months
  General Anxiety Disorder-7 (GAD-7) 12 months of follow-up
Mental health - Anxiety | 6 months
  General Anxiety Disorder-7 (GAD-7) 6 months of follow-up
Diabetes related stress | 12 months
  Problem Areas in Diabetes-5 (PAID-5) at 12 months of follow-up
Mental health - Depression | 6 months
  Patient Health Questionnaire-9 (PHQ-9) at 6 months of follow-up
Prescriptions of psychopharmacological medications | 12 months
  Prescriptions of psychopharmacological medications during one year after start of patient-inclusion. Register-based.
Medication adherence | Baseline and 12 months
  Changes in medication adherence to antidiabetic drugs and statins
Lipid profile | Baseline and 12 months
  Changes in lipid profile (from blod samples)
Blood pressure | Baseline and 12 months
  Changes in blod pressure
Smoking status | Baseline and 12 months
  Changes in smoking status
Use of health care services | Baseline and 12 months
  Changes in use of health care services including any contacts to general practice, out-of-hours medical service, cardiovascular readmissions and all cause hospitalizations
Health literacy | Baseline
  Data on health literacy will be collected at baseline using the HLSAC instrument (Health Literacy for School-Aged Children), which allows the calculation of a health literacy summary score used to examine health literacy levels. HLSAC is currently being validated among adults. The summary score is between 10-40 points: 10-25 points indicates low health literacy, 26-35 points indicates moderate health literacy, 26-40 points indicates high health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Research unit for general practice, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sojbjerg A, Mygind A, Rasmussen SE, Christensen B, Pedersen AF, Maindal HT, Burau V, Christensen KS. Improving mental health in chronic care in general practice: study protocol for a cluster-randomised controlled trial of the Healthy Mind intervention. Trials. 2024 Apr 23;25(1):277. doi: 10.1186/s13063-024-08115-8. PMID 38654329